Project No. BLI-1005-002 Statistical Analysis Plan for PDC-1421 **"Final"**  Protocol Version: 2.3 SAP Version: 20180626\_01

## 1. TITLE PAGE

# STATISTICAL ANALYSIS PLAN (SAP)

A Phase II Study of PDC-1421 Capsule to Evaluate the Safety and Efficacy in Patients with Major Depressive Disorder

| Protocol No.: | BLI-1005-002 |
|---|---|
| First subject first visit: | May-19-2015 |
| Last visit of the study: | Mar-18-2019 |
| Sponsor: | BioLite, Inc. |
| CRO: | Virginia Contract Research Organization Co., Ltd. 3F, No. 2, Lane 258, Ruiguang Rd., Neihu District, Taipei 114, Taiwan |
| Final | |
| Date of issue: | June-14-2019 |

# Project No. BLI-1005-002 Statistical Analysis Plan for PDC-1421

"Final"  Protocol Version: 2.3 SAP Version: 20180626\_01

## 2. TABLE OF CONTENTS

| 1. | TI | TLE PAGE | 1 |
|---|---|---|---|
| 2. | TA | ABLE OF CONTENTS | 2 |
| 3. | LI | ST OF ABBREVIATIONS AND DEFINITION OF TERMS | 4 |
| 4. | | ROTOCOL AMENDMENTS | |
| 5. | | VESTIGATIONAL PLAN | |
| э. | | | |
| | 5.1 | OBJECTIVE | |
| | 5.1.1 | Primary objective | |
| | 5.1.2 | Secondary objective | |
| | 5.2 | STUDY DESIGN | |
| | 5.2.1<br>5.2.2 | Schematic Diagram of The Study: | |
| | 5.2.2 | Flowchart of study procedures | |
| | 5.2.3 | STATISTICAL METHODS PLANNED IN THE PROTOCOL AND DETERMINATION OF SAMPLE SIZE | |
| | 5.3.1<br>5.3.2 | Populations for analysisEndpoints | |
| | 5.3.3 | Statistical Evaluation | |
| | 5.3.4 | Determination of sample size | |
| | 5.4 | CHANGES IN THE CONDUCT OF THE STUDY OR PLANNED ANALYSES | |
| 6. | | ATISTICAL EVALUATIONS | |
| | 6.1 | DATA SETS ANALYZED | 20 |
| | 6.2 | DEMOGRAPHICS AND OTHER BASELINE CHARACTERISTICS | 20 |
| | 6.2.1 | Demographic data | 20 |
| | 6.2.2 | Major Depressive Disorder History and Medical history | |
| | 6.2.3 | Concomitant medications | 21 |
| | 6.3 | STUDY TREATMENT ADMINISTRATION | 21 |
| | 6.3.1 | Treatment Compliance | 21 |
| | 6.3.2 | Extent of Exposure | 21 |
| | 6.3.3 | Mean Daily Dose | 21 |
| | 6.4 | Analysis of Efficacy | 22 |
| | 6.4.1 | Primary Efficacy Endpoint | |
| | 6.4.2 | Secondary efficacy endpoints: | 22 |
| | 6.5 | Analysis of Safety | 23 |
| | 6.5.1 | Adverse events (AEs) | 23 |
| | 6.5.2 | Serious adverse events (SAEs) | 23 |
| | 6.5.3 | Laboratory data | |
| | 6.5.4 | Physical Examination (PE) | |
| | 6.5.5 | Vital Signs | |
| | 6.5.6 | ECG | |
| | 6.5.7 | C-SSRS | |
| | 6.6 | STATISTICAL / ANALYTICAL ISSUES | |
| | 6.6.1 | Adjustments for covariates | |
| | 6.6.2<br>6.6.3 | Handling of Dropouts or Missing Data | |
| | 6.6.4 | Interim Analyses and Data Monitoring | |
| | 6.6.5 | Multiple Comparisons / Multiplicity | |
| | 6.6.6 | Use of An "Efficacy Subset" of Subjects | |
| | 6.6.7 | Active-Control Studies Intended to Show Equivalence | |
| | 6.6.8 | Examination of Subgroups | |

| | | CONFIDENTIAL | "Final" |
|---|---|---|---|
| | | Project No. BLI-1005-002 | Protocol Version: 2.3 |
| | | Statistical Analysis Plan for PDC-1421 | SAP Version: 20180626_01 |
| 6 | 5.6.9 | Relocation of Visit Data by Time Window | |
| 6 | 6.6.10 | Random effect and fixed effect when modeling | 26 |
| - | 6.6.11 | Outliers | |
| 6 | 5.6.12 | Calibration of Laboratory Data Between Centers | |
| 7. | DOCU | MENTATION OF STATISTICAL METHODS | 27 |
| 7.1 | Doo | CUMENTATION OF STATISTICAL METHODS | 27 |
| 8. | DATA | HANDLING PROCEDURE | 28 |
| 8.1 | Coi | DING SYSTEM | 28 |
| 8.2 | DAT | TA STORAGE AND ANALYSIS | 28 |
| 9. | STUD | Y SUBJECTS | 29 |
| 9.1 | DIS | POSITION OF SUBJECTS | 29 |
| 9.2 | WIT | THDRAWAL OF SUBJECTS | 29 |
| 9.3 | PRO | TOCOL DEVIATIONS | 29 |
| 10. | REFE | RENCE LIST | 30 |
| 11. | APPE | NDICES | 31 |
| 11.1 | Noi | RMAL RANGES FOR LABORATORY VARIABLES | 31 |
| 11.2 | 2 TAE | BLE OF CONTENTS (TOC) FOR TABLES, FIGURES AND LISTING | 31 |
| 11.3 | 8 Mo | CK-UP TABLES | 31 |
| 11.4 | VEF | RSION CONTROL INFORMATION OF SAP | 31 |
| 11.5 | 5 Con | NTENTS OF AMENDMENT OF SAP | 32 |
| 12 | SICN | ATHDE DACE | 3.4 |

Project No. BLI-1005-002 Statistical Analysis Plan for PDC-1421 "Final"  Protocol Version: 2.3 SAP Version: 20180626 01

### 3. LIST OF ABBREVIATIONS AND DEFINITION OF TERMS

AE Adverse event

BMI Body mass index

C.I. Confidence interval

CRF Case report form

CRO Contract research organization

DRCSU Depression Research Clinic at Stanford University

FDA Food and Drug Administration

GCP Good clinical practice

IQR Inter-quartile range

IRB Institutional review board

ITT Intent-to-treat

LCGMH Linkou Chang Gung Memorial Hospital

LOCF Last observation carried forward

PP Per-protocol

Q1 The first quantile (the 25<sup>th</sup> percentile)

Q3 The third quantile (the 75<sup>th</sup> percentile)

TSGH Tri-Service General Hospital

TVGH Taipei Veterans General Hospital

SAE Serious adverse event

SD Standard deviation

WH Wanfang Hospital

VCRO Virginia contract research organization

Project No. BLI-1005-002 Statistical Analysis Plan for PDC-1421

 NTIAL
 "Final" 

 I-1005-002
 Protocol Version: 2.3

 an for PDC-1421
 SAP Version: 20180626\_01

## 4. PROTOCOL AMENDMENTS

The version of approval protocol after enrolling the first subject was described as follow: As no patient were enrolled in Taipei City Hospital, Songde Branch, the site will not be included for analysis.

| Approved | | |
|---|---|---|
| date | Final | Amendment 01 |
| Approved (version: <pre>cuttor</pre> | | (version: <pre><pre>col version&gt;)</pre></pre> |
| by | ( control products , control ) | ( cossess process cosses ) |
| TFDA | 20150727 (Version 1.4) | 20160630 (Version 1.5) |
| CGMH-LK | 20150728 (Version 1.4) | 20160511 (Version 1.5) |
| TVGH | 20150806 (Version 1.4) | 20160706 (Version 1.5) |
| | | , |
| TFDA | 20160630 (Version 1.5) | 20160910 (Version 2.0) |
| CGMH-LK | 20160511 (Version 1.5) | 20160824 (Version 2.0) |
| TSGH | 20160802 (Version 1.5) | 20161017 (Version 2.0) |
| TVGH | 20160706 (Version 1.5) | 20161104 (Version 2.0) |
| TFDA | 20160910 (Version 2.0) | 20170517 (Version 2.1) |
| CGMH-LK | 20160824 (Version 2.0) | 20170406 (Version 2.1) |
| TSGH | 20161017 (Version 2.0) | 20170512 (version 2.1) |
| TVGH | 20161104 (Version 2.0) | 20170524 (Version 2.1) |
| WFH | 20161007 (version 2.0) | 20170411 (Version 2.1) |
| TFDA | 20170517 (Version 2.1) | 20171030 (Version 2.2) |
| CGMH-LK | 20170406 (Version 2.1) | 20171113 (Version 2.2) |
| TSGH | 20170512 (version 2.1) | 20171128 (Version 2.2) |
| WFH | 20170411 (Version 2.1) | 20170411 (Version 2.2) |
| TFDA | 20171030 (Version 2.2) | 20190218 (Version 2.3) |
| CGMH-LK | 20171113 (Version 2.2) | 20190214 (Version 2.3) |
| TVGH | 20170524 (Version 2.1) | 20190318 (Version 2.3) |
| WFH 20170411 (Version 2.2) | | 20190331 (Version 2.3) |
| FDA | 20170225 (Version 2.1) | 20180513 (Version 2.3) |
| Stanford | 20170128 (Version 2.1) | 20180503 (Version 2.3) |

This protocol amendment about the statistical analysis is consisted of the following

(compared to the final approved protocol):

| Page | Before | | Content after modification |
|---|---|---|---|
| | version: 1.4 | | Version: 1.5 |
| 2 | Primary endpoint Change in Montgomery-Åsberg Depression | 2 | Primary endpoint Change in Montgomery-Åsberg Depression |

Sponsor: BioLite, Inc.

**"Final"**  Protocol Version: 2.3

SAP Version: 20180626\_01


Project No. BLI-1005-002 Statistical Analysis Plan for PDC-1421

| Page | Before | Page | |
|---|---|---|---|
| rage | version: 1.4 | 1 age | Version: 1.5 |
| | Rating Scale (MADRS) total score | | Rating Scale (MADRS) total score from |
| | · | | ` / |
| | from baseline to week 4 compared to | | baseline to week 6 compared to placebo. |
| | placebo. | | |
| | | | Secondary endpoint |
| | Secondary endpoint | | Change in MADRS total score from |
| | • Change in Hamilton Rating Scale | | baseline to week 2 and 7. |
| | for Depression (HAM-D-17), | | • Change in Hamilton Rating Scale for |
| | Hamilton Rating Scale for Anxiety | | Depression (HAM-D-17), Hamilton |
| | (HAM-A), Depression and Somatic | | Rating Scale for Anxiety (HAM-A), |
| | Symptoms Scale (DSSS), Clinical | | Depression and Somatic Symptoms |
| | Global Impression Scale (CGI) total | | Scale (DSSS), Clinical Global |
| | score from baseline to week 2, 4 | | Impression Scale (CGI) total score |
| | and 5. | | from baseline to week 2, 4, 6 and 7. |
| | • Change in MADRS total score from | | • Percentage of partial responders |
| | baseline to week 2 and 5. | | (defined as a participant with a 25- |
| | <ul> <li>Percentage of partial responders</li> </ul> | | 50% decrease from baseline in total |
| | (defined as a participant with a 25- | | score) and responders (defined as a |
| | 50% decrease from baseline in total | | participant with $\geq 50\%$ decrease |
| | score) and responders (defined as a | | from baseline in total score) in |
| | participant with $\geq 50\%$ decrease | | MADRS by week 2, 4, 6 and 7. |
| | from baseline in total score) in | | Evaluate Safety Assessments and |
| | MADRS by week 2, 4 and 5. | | Columbia-Suicide Severity Rating |
| | • Evaluate Safety Assessments and | | Scale (C-SSRS) from screening stage |
| | Columbia-Suicide Severity Rating | | to the last visit |
| | Scale (C-SSRS) from screening | | • Difference in the mean changes of |
| | stage to the last visit | | MADRS, HAM-D-17, HAM-A, |
| | • Difference in the mean changes of | | DSSS, CGI and C-SSRS from the |
| | MADRS, HAM-D-17, HAM-A, | | baseline to week 2, 4, 6 and 7 |
| | DSSS, CGI and C-SSRS from the | | between the PDC-1421 Capsule and |
| | baseline to week 2, 4 and 5 between | | placebo groups. |
| | the PDC-1421 Capsule and placebo | | placebo groups. |
| | 1 - | | |
| | groups. | | 1 2 4 4 12 wools Panastad |
| | | | 1.2.4.4 13-week Repeated |
| | | | Dose Subchronic Toxicity Study in Pota |
| | | | Study in Rats |
| | | | To evaluate the subchronic toxicity of |
| | | | PDC-1421, four groups of rats were |
| 14 | None | 14 | administered with 0, 750, 1500 and |
| | | | 2500 mg/kg/once daily p.o. for 13 |
| | | | weeks (90 days). There are no |
| | | | treatment-related mortality, clinical |
| | | | signs of toxicity and ophthalmologic |
| | | | abnormality in the study. |
| | | | And no significant toxicity evidences in |

**"Final"**  Protocol Version: 2.3

SAP Version: 20180626\_01

# CONFIDENTIAL

Project No. BLI-1005-002 Statistical Analysis Plan for PDC-1421

| Page | Before | Page | |
|---|---|---|---|
| rage | version: 1.4 | rage | Version: 1.5 |
| | VCISIOII · 1.4 | | |
| | | | mean body weights, mean body weight |
| | | | gains and food consumption in all |
| | | | treatment groups were noted. |
| | | | In clinical pathology, no toxicity |
| | | | evidences were noted for all parameters |
| | | | (hematology, serum chemistry and |
| | | | urinalysis), no treatment-related gross |
| | | | abnormality was found at necropsy, and |
| | | | no significant toxicity evidences in |
| | | | organ weights evaluation. And the |
| | | | histopathological findings showed that |
| | | | no treatment-related changes in vehicle |
| | | | control and PDC-1421 treated groups. |
| | | | It was estimated that the NOAEL of |
| | | | PDC-1421 of the 13-week repeated dose |
| | | | toxicity study is 2500 mg/kg/day for |
| | | | both males and females. |
| | | 22 | |
| 22 | As Page 2 | 22 | As Page 2 |
| | 3.5.4 Dosing Regimen, packing and | | 3.5.4 Dosing Regimen, packing and |
| 2.4 | labeling Table 14. Summary of | 24 | labeling Table 14. Summary of |
| 24 | dosing regimen Visits of Part II | | dosing regimen Visits of Part II |
| | Biweekly for 28 days | | Biweekly for 42 days |
| | In part II, eligible subjects are | | In part II, eligible subjects are |
| | randomized into one of three treatment | | randomized into one of three treatment |
| | arms in a 1:1:1 ratio [one capsule of | | arms in a 1:1:1 ratio [one capsule of |
| | PDC-1421 Capsule and placebo thrice | | PDC-1421 Capsule and placebo thrice |
| | daily; two capsules of PDC-1421 | | daily; two capsules of PDC-1421 |
| | Capsule thrice daily; two capsules of | | Capsule thrice daily; two capsules |
| | placebo thrice daily] for 28 days. After | | of placebo thrice daily] for 42 days. |
| | the two weeks of drug administration, | | After the two weeks of drug |
| | subjects will return to the center for | | administration, subjects will return to |
| 25 | assessments then get another study | | the center for assessments then |
| 23 | drug bag for the following 14 days. | | get another study drug bag for the |
| | The biweekly clinic visits are two | | following 14 days. The biweekly clinic |
| | times and one week later after the last | | visits are three times and one week later |
| | dose for follow-up. | | after the last dose for follow-up. |
| | Investigational drug (PDC-1421 | | Investigational drug (PDC-1421) |
| | Capsule or placebo) are provided by | | Capsule or placebo) are provided by |
| | BioLite, Inc. and stored in Department | | BioLite, Inc. and stored in Department |
| | of Pharmacy, Taipei Veterans General | | of Pharmacy, Taipei Veterans General |
| | Hospital, Linkou Chang Gung | | Hospital, Linkou Chang Gung |
| | Memorial Hospital and Taipei City | | Memorial Hospital, Taipei City |

**"Final"**  Protocol Version: 2.3


Project No. BLI-1005-002 Statistical Analysis Plan for PDC-1421

| | Project No. B | | |
|---|---|---|---|
| D | Statistical Analysis | | |
| Page | Before | Page | Content after modification |
| | Hospital, Songde Branch. In part I, the | | Hospital, Songde Branch and Tri- |
| | first six subjects will take 21 packs | | Service General Hospital, Neihu Main |
| | with 21 capsules of PDC-1421 Capsule | | Facility and Tingihou Branch. In part I, |
| | and another six take 21 packs with 42 | | the first six subjects will take 21 packs |
| | capsules of PDC-1421 Capsule in | | with 21 capsules of PDC-1421 Capsule |
| | every week of trial. | | and another six take 21 packs with 42 |
| | In part II, subjects will be dispensed | | capsules of PDC-1421 Capsule |
| | with study drug per 2 weeks which are | | in every week of trial. In part II, |
| | packaged in a drug bag. A drug bag | | subjects will be dispensed with study |
| | will contain 42 packs. Depending on | | drug per 2 weeks which are packaged in |
| | the study arms, each pack may contain | | a drug bag. A drug bag will contain 42 |
| | 2 PDC-1421 Capsules, 2 placebos or 1 | | packs. Depending on the study |
| | PDC-1421 Capsule plus 1 placebo. | | arms, each pack may contain 2 PDC- |
| | Each subject will be administered | | 1421 Capsules, 2 placebos or 1 PDC- |
| | 84 packs in the end of trial. The drug | | 1421 Capsule plus 1 placebo. Each |
| | bag of investigational drug is clearly | | subject will be administered 126 packs |
| | labeled as following | | in the end of trial. |
| | | | The drug bag of investigational drug is |
| | | | clearly labeled as following |
| | 4.4.2 Subject Number Allocation | | 4.4.2 Subject Number Allocation |
| | The second digit: the site number; | | The second digit: the site number; |
| | Taipei Veterans General Hospital will | | Taipei Veterans General Hospital will be |
| | be assigned to "1", Linkou Chang | | assigned to "1", Linkou Chang Gung |
| | Gung Memorial Hospital will be | | Memorial Hospital will be assigned to |
| 32 | assigned to "2" and Taipei City | 32 | "2" and Taipei City Hospital, Songde |
| | Hospital, Songde Branch will be | | Branch will be assigned to 3", Tri- |
| | assigned to "3". | | Service General Hospital, Neihu |
| | | | Main Facility will be assigned to "4". |
| | | | Tri-Service General Hospital, Tingjhou |
| | | | Branchwill be assigned to "5". |
| | 10.4 Institutional Review Board (IRB) | | 10.4 Institutional Review Board (IRB) |
| | This study is conducted to be | | This study is conducted to be consistent |
| | consistent with the principles of the | | with the principles of the Declaration of |
| | Declaration of Helsinki and GCP. This | | Helsinki and GCP. This protocol and |
| | protocol and any supplementary | | any supplementary documents, |
| | documents, including written | | including written informed consent |
| | informed consent form, subject | | form, subject recruitment |
| 52 | recruitment advertisements and | 52 | advertisements and Investigator's |
| | Investigator's Brochure, must be | | Brochure, must be reviewed and |
| | reviewed and approved by IRB of | | approved by IRB of the |
| | the Taipei Veterans General Hospital, | | Taipei Veterans General Hospital, |
| | Linkou Chang Gung Memorial | | Linkou Chang Gung Memorial |
| | Hospital and Taipei City Hospital, | | Hospital, Taipei City Hospital, Songde |
| | Songde Branch qualified with local | | Branch and Tri-Service General |

Sponsor: BioLite, Inc.

Project No. BLI-100
Statistical Analysis Plan fo

| IAI | | "Final" |
|-----|------------------------------|--------------------------|
| 005 | -002 | Protocol Version: 2.3 |
| for | PDC-1421 | SAP Version: 20180626_01 |
| ge | e Content after modification | |

| Page | | Befor | re | | | Page | Content after modification |
|---|---|---|---|---|---|---|---|
| | | version | : 1.4 | | | | Version: 1.5 |
| | legal<br>initiati | prescriptions on | prior | to | study | | Hospital qualified with local legal prescriptions prior to study initiation |

| Page Before version: 1.4 Primary endpoint | Page | Version: 1.5 |
|---|---|---|
| Change in Montgomery Depression Rating Scale (MADRS) total from baseline to week 4 complacebo. Secondary endpoint Change in Hamilton Rating for Depression (HAM Hamilton Rating Scale for (HAM-A), Depression and Symptoms Scale (DSSS), Global Impression Scale (CC score from baseline to we and 5. Change in MADRS total score baseline to week 2 and 5. Percentage of partial respond (defined as a participant with 50% decrease from baseline score) and responders (define participant with ≥ 50% of from baseline in total score) and from the from | g Scale I-D-17), Anxiety Somatic Clinical GI) total ek 2, 4 re from 2 lers h a 25- in total led as a lecrease ore) in s and lecrease ore) in ges of IAM-A, rom the between | Primary endpoint Change in Montgomery-Åsberg Depression Rating Scale (MADRS) total score from baseline to week 6 compared to placebo. Secondary endpoint Change in MADRS total score from baseline to week 2 and 7. Change in Hamilton Rating Scale for Depression (HAM-D-17), Hamilton Rating Scale for Anxiety (HAM-A), Depression and Somatic Symptoms Scale (DSSS), Clinical Global Impression Scale (CGI) total score from baseline to week 2, 4, 6 and 7. Percentage of partial responders (defined as a participant with a 25- 50% decrease from baseline in total score) and responders (defined as a participant with ≥ 50% decrease from baseline in total score) in MADRS by week 2, 4, 6 and 7. Evaluate Safety Assessments and Columbia-Suicide Severity Rating Scale (C-SSRS) from screening stage to the last visit Difference in the mean changes of MADRS, HAM-D-17, HAM-A, DSSS, CGI and C-SSRS from the baseline to week 2, 4, 6 and 7 between the PDC-1421 Capsule and placebo groups. |

Project No. BLI-1005-002 Statistical Analysis Plan for PDC-1421

**"Final"**  Protocol Version: 2.3 SAP Version: 20180626 01

| D | Statistical Analysis | | - |
|---|---|---|---|
| Page | Before | Page | Content after modification |
| 14 | None | 14 | 1.2.4.4 13-week Repeated Dose Subchronic Toxicity Study in Rats To evaluate the subchronic toxicity of PDC-1421, four groups of rats were administered with 0, 750, 1500 and 2500 mg/kg/once daily p.o. for 13 weeks (90 days). There are no treatment-related mortality, clinical signs of toxicity and ophthalmologic abnormality in the study. And no significant toxicity evidences in mean body weights, mean body weight gains and food consumption in all treatment groups were noted. In clinical pathology, no toxicity evidences were noted for all parameters (hematology, serum chemistry and urinalysis), no treatment-related gross abnormality was found at necropsy, and no significant toxicity evidences in organ weights evaluation. And the histopathological findings showed that no treatment-related changes in vehicle control and PDC-1421 treated groups. It was estimated that the NOAEL of PDC-1421 of the 13-week repeated dose toxicity study is 2500 mg/kg/day for both males and females. |
| 22 | As Page 2 | 22 | As Page 2 |
| 24 | 3.5.4 Dosing Regimen, packing and labeling Table 14. Summary of dosing regimen Visits of Part II Biweekly for 28 days | 24 | 3.5.4 Dosing Regimen, packing and labeling Table 14. Summary of dosing regimen Visits of Part II Biweekly for 42 days |
| 25 | In part II, eligible subjects are randomized into one of three treatment arms in a 1:1:1 ratio [one capsule of PDC-1421 Capsule and placebo thrice daily; two capsules of PDC-1421 Capsule thrice daily; two capsules of placebo thrice daily] for 28 days. After the two weeks of drug administration, | | In part II, eligible subjects are randomized into one of three treatment arms in a 1:1:1 ratio [one capsule of PDC-1421 Capsule and placebo thrice daily; two capsules of PDC-1421 Capsule thrice daily; two capsules of placebo thrice daily] for 42 days. After the two weeks of drug |

**"Final"**  Protocol Version: 2.3

SAP Version: 20180626\_01


Project No. BLI-1005-002 Statistical Analysis Plan for PDC-1421

| Page | Before | Page | Content after modification |
|---|---|---|---|
| 8 | version: 1.4 | 8- | Version: 1.5 |
| | subjects will return to the center for | | administration, subjects will return to |
| | assessments then get another study | | the center for assessments then |
| | drug bag for the following 14 days. | | get another study drug bag for the |
| | The biweekly clinic visits are two | | following 14 days. The biweekly clinic |
| | times and one week later after the last | | visits are three times and one week later |
| | dose for follow-up. | | after the last dose for follow-up. |
| | Investigational drug (PDC-1421 | | Investigational drug (PDC-1421) |
| | Capsule or placebo) are provided by | | Capsule or placebo) are provided by |
| | BioLite, Inc. and stored in Department | | BioLite, Inc. and stored in Department |
| | of Pharmacy, Taipei Veterans General | | of Pharmacy, Taipei Veterans General |
| | Hospital, Linkou Chang Gung | | Hospital, Linkou Chang Gung |
| | Memorial Hospital and Taipei City | | Memorial Hospital, Taipei City |
| | Hospital, Songde Branch. In part I, the | | Hospital, Songde Branch and Tri- |
| | first six subjects will take 21 packs | | Service General Hospital, Neihu Main |
| | with 21 capsules of PDC-1421 Capsule | | Facility and Tingjhou Branch. In part I, |
| | and another six take 21 packs with 42 | | the first six subjects will take 21 packs |
| | capsules of PDC-1421 Capsule in | | with 21 capsules of PDC-1421 Capsule |
| | every week of trial. | | and another six take 21 packs with 42 |
| | In part II, subjects will be dispensed | | capsules of PDC-1421 Capsule |
| | with study drug per 2 weeks which are | | in every week of trial. In part II, |
| | packaged in a drug bag. A drug bag | | subjects will be dispensed with study |
| | will contain 42 packs. Depending on | | drug per 2 weeks which are packaged in |
| | the study arms, each pack may contain | | a drug bag. A drug bag will contain 42 |
| | 2 PDC-1421 Capsules, 2 placebos or 1 | | packs. Depending on the study |
| | PDC-1421 Capsule plus 1 placebo. | | arms, each pack may contain 2 PDC- |
| | Each subject will be administered | | 1421 Capsules, 2 placebos or 1 PDC- |
| | 84 packs in the end of trial. The drug | | 1421 Capsule plus 1 placebo. Each |
| | bag of investigational drug is clearly | | subject will be administered 126 packs |
| | labeled as following | | in the end of trial. |
| | | | The drug bag of investigational drug is |
| | | | clearly labeled as following |
| | 4.4.2 Subject Number Allocation | | 4.4.2 Subject Number Allocation |
| | The second digit: the site number; | | The second digit: the site number; |
| | Taipei Veterans General Hospital will | | Taipei Veterans General Hospital will be |
| | be assigned to "1", Linkou Chang | | assigned to "1", Linkou Chang Gung |
| | Gung Memorial Hospital will be | | Memorial Hospital will be assigned to |
| 32 | assigned to "2" and Taipei City | 32 | "2" and Taipei City Hospital, Songde |
| | Hospital, Songde Branch will be | | Branch will be assigned to 3", Tri- |
| | assigned to "3". | | Service General Hospital, Neihu |
| | | | Main Facility will be assigned to "4". |
| | | | Tri-Service General Hospital, Tingjhou |
| | | | Branchwill be assigned to "5". |

Project No. BLI-1005-002 Statistical Analysis Plan for PDC-1421

"Final"  Protocol Version: 2.3 SAP Version: 20180626\_01

| Page | Before | Page | Content after modification |
|---|---|---|---|
| | 10.4 Institutional Review Board (IRB) | | 10.4 Institutional Review Board (IRB) |
| | This study is conducted to be | | This study is conducted to be consistent |
| | consistent with the principles of the | | with the principles of the Declaration of |
| | Declaration of Helsinki and GCP. This | | Helsinki and GCP. This protocol and |
| | protocol and any supplementary | | any supplementary documents, |
| | documents, including written | | including written informed consent |
| | informed consent form, subject | | form, subject recruitment |
| 17/ | recruitment advertisements and | 52 | advertisements and Investigator's |
| | investigator's Brochure, must be | 32 | Brochure, must be reviewed and |
| | reviewed and approved by IRB of | | approved by IRB of the |
| | the Taipei Veterans General Hospital, | | Taipei Veterans General Hospital, |
| | Linkou Chang Gung Memorial | | Linkou Chang Gung Memorial |
| | Hospital and Taipei City Hospital, | | Hospital, Taipei City Hospital, Songde |
| | Songde Branch qualified with local | | Branch and Tri-Service General |
| | legal prescriptions prior to study | | Hospital qualified with local legal |
| | initiation | | prescriptions prior to study initiation |

| Page | Before | Page | Content after modification |
|---|---|---|---|
| | version: 1.5 | | Version: 2.0 |
| 32 | version: 1.5 4.4.2 Subject Number Allocation The second digit: the site number; Taipei Veterans General Hospital will be assigned to "1", Linkou Chang Gung Memorial Hospital will be assigned to "2" and Taipei City Hospital, Songde Branch will be assigned to "3", Tri-Service General Hospital, Neihu Main Facility will be assigned to "4". Tri-Service General Hospital, Tingjhou Branchwill be | 32 | 4.4.2 Subject Number Allocation The second digit: the site number. |
| | assigned to "5". | | |

| Page | Before | Page | Content after modification |
|---|---|---|---|
| | version: 2.1 | | Version: 2.2 |
| | 3.1 General Design | | 3.1 General Design |
| | The targeted population of this study is | | The targeted population of this study is |
| 21 | 72 subjects who met the per-protocol | 21 | 72 subjects who met the intent-to-treat |
| | basis, in which 12 are assigned to part | | (ITT) basis, in which 12 are assigned to |
| | I, 60 are assigned to part II. | | part I, 60 are assigned to part II. |

Project No. BLI-1005-002 Statistical Analysis Plan for PDC-1421

"Final"  Protocol Version: 2.3 SAP Version: 20180626\_01

| Page | Before | Page | Content after modification |
|---|---|---|---|
| | 8.1 Sample Size Determination | | 8.1 Sample Size Determination |
| 48 | Based on our study design, it is | 10 | Based on our study design, it is planned |
| 48 | Based on our study design, it is planned to enroll 60 subjects who met | | to enroll 60 subjects who met the intent- |
| | the per-protocol basis. | | to-treat (ITT) basis. |

| Page | Before | | Content after modification |
|---|---|---|---|
| | version: 2.2 | | Version: 2.3 |
| | | | Percentage of partial responders |
| | The total score is used to define | | (defined as a participant with a 25-50% |
| 42 | treatment response (≥40% reduction | 12 | decrease from baseline in total score) |
| 42 | from baseline) and partial response | | and responders (defined as a participant |
| | (20-39% reduction from baseline). | | with $\geq 50\%$ decrease from baseline in |
| | | | total score. |

Project No. BLI-1005-002 Statistical Analysis Plan for PDC-1421 "Final"  Protocol Version: 2.3 SAP Version: 20180626 01

### 5. INVESTIGATIONAL PLAN

### 5.1 Objective

### 5.1.1 Primary objective

The primary objective of this trial was to determine the effective doses and treatment period of PDC-1421 Capsule in subjects with MDD.

## 5.1.2 Secondary objective

To evaluate the safety of PDC-1421 Capsule in subjects receiving PDC-1421 at various dose levels .

# 5.2 Study Design

The screening phase is intended for diagnosing and assessing the patient for possible inclusion in the study and for providing an adequate washout period. The following study will be conducted in two parts. The targeted population of this study is 72 subjects who met the intent-to-treat (ITT) basis, in which 12 are assigned to part I, 60 are assigned to part II. Part I is an open-label study, multiple center and dose escalation evaluation in twelve patients. Six subjects each will be evaluated for any safety concerns at 1 or 2 capsules TID dose for 28 days, sequentially. Each of them will be assessed twice in the first week after administration of PDC-1421 Capsules and once a week in the following treatment. Part II is a randomized, double-blind, placebo-controlled, parallel-group study. 60 subjects will be randomly assigned on a 1:1:1 basis to one of the three treatment arms (1 PDC-1421 Capsule plus 1 placebo TID, 2 PDC-1421 Capsule TID, 2 placebo TID) for 6 weeks (42 days) and evaluated the safety and efficacy every two weeks during the treatment period. The performance of PDC-1421 Capsule on MDD subjects will provide us with valuable information for our next phase of the study.

Sponsor: BioLite, Inc.

Project No. BLI-1005-002 Statistical Analysis Plan for PDC-1421 "Final"  Protocol Version: 2.3 SAP Version: 20180626 01

## 5.2.1 Schematic Diagram of The Study:

Part I.



<sup>\*</sup> Subjects are assessed once between visit 2 and 4

□ Checkpoints

Part II.



Sponsor: BioLite, Inc.

Project No. BLI-1005-002 Statistical Analysis Plan for PDC-1421 "Final"  Protocol Version: 2.3 SAP Version: 20180626 01

### 5.2.2 Study Medication Administration

In part I, six subjects each will take 1 or 2 capsules thrice daily for 28 days, sequentially. Subjects are assessed twice in the first week after drug administration and they will receive the study drug bag for the following 7 days every week. In part II, eligible subjects are randomized into one of three treatment arms in a 1:1:1 ratio (one capsule of PDC-1421 Capsule and placebo thrice daily; two capsules of PDC-1421 Capsule thrice daily; two capsules of placebo thrice daily) for 42 days. After the two weeks of drug administration, subjects will return to the center for assessments then get another study drug bag for the following 14 days. The biweekly clinic visits are three times and one week later after the last dose for follow-up.

## 5.2.3 Flowchart of study procedures

Part I-schedule of assessments

\*On  $\pm 2$  days.

\*V3 (Week 1/2) only can be conducted in Day 3 or Day 4.

| | Screening | | Tı | eatme | nt Peri | od | | Follow-up |
|---|---|---|---|---|---|---|---|---|
| Visit | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 |
| *Week | -2 to -1 ~0 | 0 | 1/2 | 1 | 2 | 3 | 4 | 5 |
| Informed consent | • | | | | | | | |
| Subject information | • | | | | | | | |
| Medical history | • | • | | | | | | |
| DSM-IV-TR | • | | | | | | | |
| HAM-D-17 | • | • | | • | • | • | • | • |
| CGI | • | • | | • | • | • | • | • |
| MADRS | • | • | | • | • | • | • | • |
| DSSS | • | • | | • | • | • | • | • |
| HAM-A | • | • | | • | • | • | • | • |
| C-SSRS | • | • | • | • | • | • | • | • |
| Concomitant | • | • | • | • | • | • | • | • |
| medication | | | | | | | | |
| Physical | • | • | • | • | • | • | • | • |
| examination | | | | | | | | |
| Vital sign | • | • | • | • | • | • | • | • |
| ECG | • | • | • | • | • | • | • | • |
| Laboratory | | | | | | | | |
| examination | | | | | | | | |
| Drug screen | • | | | | | | | |
| Pregnancy test | • | | | | | | | • |
| Hematology | • | • | | | • | | • | • |
| Blood chemistry | • | • | | | • | | • | • |
| Eligibility evaluation | • | | | | | | | |
| Drug accountability | | • | • | • | • | • | • | |
| AE/SAE evaluation | | | • | • | • | • | • | • |

Sponsor: BioLite, Inc.

"Final" 

#### **CONFIDENTIAL**

Project No. BLI-1005-002 Statistical Analysis Plan for PDC-1421

Protocol Version: 2.3 SAP Version: 20180626 01

Part II-schedule of assessments

\*\* If the interval of visit 1 and visit 2 is within 7 days, Hematology and Blood chemistry test of visit 2 can be skipped.

| | Screening | | Treatm | eut Peri | od | Follow-up |
|---|---|---|---|---|---|---|
| Visit | 1 | 2 | 3 | 4 | 5 | 6 |
| *Week | -2 to -1 ~ 0 | 0 | 2 | 4 | 6 | 7 |
| Informed consent | • | | | | | |
| Subject information | • | | | | | |
| Medical history | • | • | | | | |
| DSM-IV-TR | • | | | | | |
| HAM-D-17 | • | • | • | • | • | • |
| CGI | • | • | ٠ | ٠ | ٠ | ٠ |
| MADRS | • | • | ٠ | ٠ | ٠ | • |
| DSSS | • | • | ٠ | ٠ | ٠ | • |
| HAM-A | • | • | • | • | • | • |
| C-SSRS | • | • | • | • | • | • |
| Concomitant | • | • | • | • | • | • |
| medication | | | | | | |
| Physical examination | • | • | • | • | • | • |
| Vital sign | • | • | • | • | • | • |
| ECG | • | • | • | • | • | • |
| Laboratory | | | | | | |
| examination | | | | | | |
| Drug screen | • | | | | | |
| Pregnancy test | • | | | | | • |
| Hematology | • | •" | • | • | ٠ | • |
| Blood chemistry | • | •" | • | • | • | • |
| Eligibility evaluation | • | | | | | |
| Drug accountability | | • | • | • | • | |
| AE/SAE evaluation | | | • | • | • | • |

#### 5.3 Statistical Methods Planned in the Protocol and Determination of Sample Size

#### 5.3.1 Populations for analysis

The efficacy measures are conducted on the per-protocol (PP) and intent-to-treat (ITT) basis. The per protocol will be defined as (1) The drug compliance is at least 80% (2) Subjects have completed data to determine the primary endpoint. (3) Subjects cannot have protocol deviation. The protocol deviation will be defined as (1) Inclusion or exclusion criteria not satisfied. (2) Not permitted concomitant medications (3) Wrong randomized treatment prescribed. An intent-to-treat (ITT) basis will be defined as the data are analyzed by the treatment groups to which the randomized patients who take at least one dose of study medication and have any post-baseline safety data collected.

The safety measures are conducted on the ITT basis.

#### 5.3.2 **Endpoints**

## **Primary endpoint:**

Sponsor: BioLite, Inc.

<sup>\*</sup>On  $\pm 2$  days.

Project No. BLI-1005-002 Statistical Analysis Plan for PDC-1421 "Final"  Protocol Version: 2.3 SAP Version: 20180626 01

In part II, the primary endpoint is the change of Montgomery-Å sberg Depression Rating Scale (MADRS) total score from baseline to Week 6 compared to placebo.

## Secondary endpoints are:

- MADRS total score—change from baseline to week 2 and 7
- HAM-D-17, CGI, DSSS and HAM-A—change from baseline to week 2, 4, 6 and 7
- Percentage of partial responders and responders (defined as participants with a 25-50% decrease and a  $\geq$  50% decrease from baseline in total score, respectively) in MADRS total score by Week 2, 4, 6 and 7
- Difference in the mean changes of MADRS, HAM-D-17, HAM-A,DSSS, CGI and C-SSRS from baseline to week 2, 4, 6 and 7 between PDC-1421 Capsule and placebo groups.

## Safety endpoints:

- physical examination
- vital signs
- laboratory data (blood chemistry)
- FCG
- Columbia-Suicide Severity Scale (C-SSRS)
- Incidence of AE/SAE

#### 5.3.3 Statistical Evaluation

Simple descriptive statistics with 95% confidence interval will be performed with data collected in this study wherever applicable. Treatment effects are evaluated based on 2-sided test with a 0.05 significant level. All data shall be tabulated and presented in the study report. The descriptive statistics will be provided. The safety and efficacy data will be analyzed using the non-parametric method.

### 5.3.3.1 Primary analysis methods

The efficacy and safety information recorded on CRF will be summarized by tables presented in frequency and percentage for categorical variables, in mean with SD as well as median with the minimum and maximum for continuous variables. The comparison between three groups will be analyzed by nonparametric method as appropriate. All adverse events will be summarized with coding term, severity, relationship to study drug by frequency tables with the counts and percentage. In addition, serious adverse events will be listed with event narration.

### 5.3.4 Determination of sample size

In part I, six subjects each will be evaluated for safety and efficacy assessments at 1 or 2 capsules TID dose for 28 days, sequentially.

Sponsor: BioLite, Inc.

Project No. BLI-1005-002 Statistical Analysis Plan for PDC-1421 "Final"  Protocol Version: 2.3

SAP Version: 20180626\_01

In part II, this is a small proof-of-concept study to evaluate 2 doses of PDC-1421 and placebo in the treatment of major depressive disorder. Based on our study design, it is planned to enroll 60 subjects who met the intent-to-treat (ITT) basis.

# 5.4 Changes in the Conduct of the Study or Planned Analyses

All the statistical analysis will follow protocolized statistical contents.

Project No. BLI-1005-002 Statistical Analysis Plan for PDC-1421

### "Final"  Protocol Version: 2.3 SAP Version: 20180626 01

### 6. STATISTICAL EVALUATIONS

The statistical objective of this study is to assess the safety and efficacy profiles in three groups - 1 PDC-1421 capsule plus 1 placebo, 2 PDC-1421 Capsule, and 2 placebos.

### 6.1 Data Sets Analyzed

Two study populations are intention-to-treat (ITT) population and per-protocol (PP) populations which are defined in section 5.3.1.

The efficacy evaluations will be performed on both of the ITT and PP datasets while the safety evaluations will be performed on the ITT dataset. The primary conclusion will be made for the primary endpoint on the ITT population

Demographic and baseline (Visit 2) characteristics will be performed on the ITT population.

Sample size, mean, 95% confidence interval of mean, median, standard deviation, interquartile range, maximum and minimum will be summarized for continuous variables. For categorical variables, the frequency and percentage will be provided.

### 6.2 Demographics and Other Baseline Characteristics

Demography and baseline characteristics will be summarized in descriptive statistics and listed by part, center and treatment.

### 6.2.1 Demographic data

Demographic variables including age(year), height (cm), weight (kg) and BMI (kg/m²) will be summarized. Subjects' gender will be tabulated.

Age (years) = integer of (date of initial visit – date of birth) / 365.25

BMI  $(Kg/m^2) = (weight) / (height)^2$  rounds to one decimal place

## 6.2.2 Major Depressive Disorder History and Medical history

Frequency table of Diagnosis and Statistical Manual of Mental Disorders-IV, text revision (DSM-IV-TR) will be presented.

Frequency table of subject with medical history and current medical condition will be presented.

Sponsor: BioLite, Inc.

Project No. BLI-1005-002 Statistical Analysis Plan for PDC-1421 **"Final"**  Protocol Version: 2.3

SAP Version: 20180626 01

General medical history will be presented in incidence table and listed for each subject. Ongoing medical conditions will be presented separately from the cured diseases.

#### 6.2.3 Concomitant medications

Frequency table of subjects with pre-treatment and concomitant medications will be presented. WHO Drug Dictionary will be applied.

Pre-treatment medications are the medications taken before the first dosing of study drug, while concomitant medications are those taken during the treatment duration (from first dosing date of study drug to the day before exiting from study).

#### 6.3 **Study Treatment Administration**

#### 6.3.1 Treatment Compliance

Subjects' compliance (%) during the treatment period will be tabulated by part, center, and treatment and calculated according to the following formula:

= 100\* Number of study medication actually took during the extent of exposure Number of study medication should be taken during the extent of exposure (#)

# = (number of study medication should be taken per day) \* (extent of exposure, section 6.3.2)

#### 6.3.2 Extent of Exposure

Extent of exposure (days) = date of last drug taken - date of first drug taken + 1

If the date of first drug taken is not available, the date when the drug was firstly dispensed will be used for calculation.

If the date of last drug taken is not available, the date will be replaced with that of the last drug return, previous drug taken, or previous drug return in order.

#### 6.3.3 Mean Daily Dose

Descriptive statistics of mean daily dose of the test drug will be presented by part, center, and treatment.

> Number of study medication taken Mean daily dose = Extent of exposure (section 6.3.2)

Sponsor: BioLite, Inc.

Project No. BLI-1005-002 Statistical Analysis Plan for PDC-1421 "Final"  Protocol Version: 2.3 SAP Version: 20180626 01

### 6.4 Analysis of Efficacy

Results of efficacy will be presented with descriptive statistics (i.e. sample size, number of missing data, mean, 95% confidence interval of mean, median, standard deviation, interquartile range, maximum and minimum) for continuous parameters by part, visit, and treatment. Line charts of all efficacy outcomes will be generated and presented as mean and standard deviation.

## 6.4.1 Primary Efficacy Endpoint

In part II study, the primary endpoint is the net change of the MADRS total score at the 6th week after treatment (Mean MADRS total score at week 6 – Mean MADRS total score at baseline [Visit 2]).

Kruskal-Wallis test will be implemented to test the group difference.

The primary hypothesis will be:

H<sub>0</sub>: The mean ranks of the groups are the same

H<sub>a</sub>: The mean ranks of the groups are not the same

One a significant treatment effect is found, Wilcoxon rank sum test with Holm procedure will then be performed for comparisons between two treatment groups and the placebo group. The treatment group will be declared superior if null hypothesis is rejected and  $\mu_{t1}$  and/or  $\mu_{t2}$  is greater than  $\mu_p$ .

### 6.4.2 Secondary efficacy endpoints:

In the part II study, change from baseline in MADRS at week 2/4/7, along with net changes in HAM-D-17, HAM-A, DSSS, and CGI at week 2/4/6/7 are the secondary endpoints. Also, group differences in net changes of the MADRS, CGI, HAM-D-17, HAM-A, and DSSS at the 2<sup>nd</sup>, 4<sup>th</sup>, 6<sup>th</sup>, and 7<sup>th</sup> week are the secondary efficacy endpoints. For the results with regard to MADRS and HAM-D-17, the summary of all sites in Taiwan will also be provided to contrast with the one in America.

Descriptive statistics for original and changes from baseline will be display by part, center, visit and treatment. As for the group difference, it will be examined by Kruskal-Wallis test. A significant treatment effect will be claimed after the Wilcoxon rank sum test for post-hoc tests.

In addition to the treatment difference, the effect of different product batches (or batch number)- the first batch and the second batch, on MADRS will also be examined. Drugs with batch number of "HDP-045A-040327" and placebos with batch number of "HDP-045C-040327" are classified into the first batch of product. The batch numbers included in the

Sponsor: BioLite, Inc.

Project No. BLI-1005-002 Statistical Analysis Plan for PDC-1421 "Final"  Protocol Version: 2.3 SAP Version: 20180626 01

second batch are "HDP-045A-070119" for PDC-1421 and "HDP-045C-070119" for placebo. Subjects with baseline visit later than 2018/02/13, or those who were enrolled before 2018/02/13 and got drugs after 2018/03/15 will be classified into the subgroup of the second batch.

The responder and partial responder is defined by the net change in total score of MADRS (responders are defined as participants with a  $\geq 50\%$  decrease in total score from baseline; partial responders are defined as participants with at least 25% and no more than 50% decrease in total score from baseline). The percentage difference between treatment groups will be examined by Cochran-Mantel-Haenszel test.

The same definitions of partial responder will be used for HAM-D-17. The difference between the treatment will be compared with Cochran-Mantel-Haenszel test as well.

All statistical tests used will be two-tailed with  $\alpha = 0.05$ .

### 6.5 Analysis of Safety

### 6.5.1 Adverse events (AEs)

The coding system used will be the Medical Dictionary for Regulatory Activities (MedDRA).

Pre-treatment AE is the AE onset before the first dosing of study drug, while treatmentemergent AE is the one onset after the first dosing of study drug. Pre-treatment AE and treatment emergent AE will be analyzed separately.

Frequency table of subjects with pre-treatment AE (PTAE) and treatment emergent AE (TEAE) will be presented by part, center and treatment.

For TEAE, adverse event incidents will also be summarized descriptively by system organ class and preferred term using MedDRA. If more than one type of event occurred within a system organ class/ preferred term for the subject, the subject is counted only once for each system organ class/ preferred term.

For TEAE, incidence tables of severity, action taken, relationship to study drug, outcome and serious AE or not will be presented by part, center, preferred term and treatment.

The frequency distribution of severity, action taken, relationship to study drug, and outcome of all AE events will be presented by part, center, and treatment.

### 6.5.2 Serious adverse events (SAEs)

Incidence of serious adverse event will be tabulated. Serious adverse events incidents will be summarized descriptively by part, center, system organ class/ preferred term, and treatment group.

Project No. BLI-1005-002 Statistical Analysis Plan for PDC-1421 "Final"  Protocol Version: 2.3 SAP Version: 20180626 01

## 6.5.3 Laboratory data

Descriptive statistics of original data and net changes in hematology and biochemistry data will be presented by part, center, visit, and treatment.

Results of clinical significance with regard to laboratory data will be summarized with frequency and percentage.

### 6.5.4 Physical Examination (PE)

Incidence table including umber and percentage of patient with abnormal PE will be tabulated by part, center, visit, and treatment for each body system.

The corresponding body system will be analyzed and reported using a transition table. The type of transition includes no change, change to normal, change to non-clinical significance, (NCS), change to clinical significance (CS) for each body system from baseline (Visit 2).

### 6.5.5 Vital Signs

Descriptive statistics of net changes in vital signs including systolic and diastolic blood pressure, heart rate and body temperature will be presented by part, center, visit, and treatment.

Results of clinical significance with regard to vital sign will be summarized with frequency and percentage.

#### 6.5.6 ECG

Frequency table and change in ECG result will be summarized by part, center, visit and treatment. The transition of ECG is define as following 4 groups: no change, change to normal, change to non-clinical significance, (NCS), change to clinical significance (CS).

#### 6.5.7 C-SSRS

Results of C-SSRS will be presented by part, center, visit, and treatment. The baseline of C-SSRS was set at screening visit (Visit 1).

The analysis for C-SSRS will follow the official guidance "Columbia-Suicide Severity Rating Scale - Scoring and Data Analysis Guide." The 10 categories will be defined according to 10 binary responses (yes/no) on the C-SSRS, which are:

Category 1 – Wish to be Dead

Category 2 – Non-specific Active Suicidal Thoughts

Category 3 – Active Suicidal Ideation with Any Methods (Not Plan) without Intent to Act

Category 4 – Active Suicidal Ideation with Some Intent to Act, without Specific Plan

Sponsor: BioLite, Inc.

**"Final"** 

Protocol Version: 2.3

#### CONFIDENTIAL

Project No. BLI-1005-002 Statistical Analysis Plan for PDC-1421 SAP Version: 20180626 01

Category 5 – Active Suicidal Ideation with Specific Plan and Intent

Category 6 – Preparatory Acts or Behavior

Category 7 – Aborted Attempt

Category 8 – Interrupted Attempt

Category 9 – Actual Attempt (non-fatal)

Category 10 – Completed Suicide

Suicidal ideation is identified if the total score of the five suicidal ideation questions (Categories 1-5)>0. Suicidal behavior is identified if the total score of the five suicidal behavior questions (Categories 6-10)>0. Suicidal ideation or behavior is identified if the total score of the ten suicidal ideation and behavior questions (Categories 1-10)>0.

Changes of suicidal ideation, suicidal behavior, and suicidal ideation or behavior from baseline during treatment will be summarized in a shift-table by visit, center and treatment.

#### 6.6 **Statistical / Analytical Issues**

#### 6.6.1 Adjustments for covariates

No adjustment for covariates will be performed in this study.

#### 6.6.2 Handling of Dropouts or Missing Data

Missing data caused by premature termination will be utilized the last observation carried forward (LOCF). However, the LOCF method will only be applied to data on efficacy. No imputation will be done for safety data.

#### 6.6.3 Interim Analyses and Data Monitoring

No interim analysis was planned.

#### 6.6.4 Multicenter Studies

This is a multi-center study, which was conducted in the Depression Research Clinic at Stanford University, Tri-Service General Hospital, Taipei Veterans General Hospital, Linkou Chang Gung Memorial Hospital, Taipei City Hospital, Songde Branch, and Wanfang Hospital. All results will be listed by center.

#### 6.6.5 Multiple Comparisons / Multiplicity

The Holm procedure will be carried out for the post-hoc test of the primary endpoint.

#### 6.6.6 Use of An "Efficacy Subset" of Subjects

All analyzed populations were defined in section 5.3.1; no other population will be utilized in statistical analyses.

Sponsor: BioLite, Inc.

Project No. BLI-1005-002 Statistical Analysis Plan for PDC-1421 "Final"  Protocol Version: 2.3 SAP Version: 20180626 01

## 6.6.7 Active-Control Studies Intended to Show Equivalence

Not applicable

### 6.6.8 Examination of Subgroups

No subgroup analysis was conducted in the study. All center data will be pooled together for analyses of efficacy endpoint.

## 6.6.9 Relocation of Visit Data by Time Window

Subject with visit relocation are listed in table below:

| Obs | Subject number | Visit on CRF | Real date of visit | Reallocated visit | Decision from sponsor |
|---|---|---|---|---|---|
| 8 | 11-07-07 | 8 | 2016/04/11 | 7 | 8 |
| 14 | 21-07-08 | 6 | 2017/04/12 | 4 | 4 |
| 20 | 21-08-07 | 6 | 2017/05/03 | 5 | 5 |
| 26 | 21-10-10 | 6 | 2017/04/18 | 3 | 4 |
| 32 | 21-19-19 | 6 | 2017/12/06 | 3 | 3 |
| 38 | 21-26-25 | 6 | 2018/06/04 | 3 | 3 |
| 44 | 21-27-26 | 6 | 2018/12/01 | 999 | 3 |
| 48 | 22-03-02 | 6 | 2017/01/11 | 3 | 3 |
| 53 | 22-04-03 | 5 | 2017/02/15 | 6 | 5 |
| 59 | 22-06-05 | 6 | 2017/04/25 | 4 | 4 |
| 64 | 27-03-02 | 5 | 2018/08/07 | 6 | 5 |

<sup>\* 999=</sup> cannot be determined

## 6.6.10 Random effect and fixed effect when modeling

Not applicable

### **6.6.11** *Outliers*

Outliers will not be excluded for and some extreme values will be excluded from this study.

## 6.6.12 Calibration of Laboratory Data Between Centers

Units of continuous laboratory data will be unified; the ones used in a plurality of center will be the standard.

Sponsor: BioLite, Inc.

Project No. BLI-1005-002 Statistical Analysis Plan for PDC-1421 **"Final"**  Protocol Version: 2.3 SAP Version: 20180626 01

## 7. DOCUMENTATION OF STATISTICAL METHODS

## 7.1 Documentation of Statistical Methods

Following SAS procedures will be applied for statistical methods mentioned in Chapter 6.

| SAS | Statistical Analysis | Comment |
|---|---|---|
| procedure | Method | |
| Freq | Frequency table | |
| | Cochran-Mantel- | Test of association between variables by controlling |
| | Haenszel Test | for multiple centers |
| Sgplot | Graph | |
| NPAR1WAY | Kruskal-Wallis test | To test group difference of continuous variables |
| | Wilcoxon rank sum test | Post-hoc test |
| MULTTEST | Holm's Procedure | Significant level control for Multiplicity |
| MEANS | Descriptive Statistics | Means, SD, Min, Max, Med, IQR, P1, P3 |

<sup>\*</sup>Center effect will be incorporated in only when degree of freedom is sufficient.

Sponsor: BioLite, Inc.

Project No. BLI-1005-002 Statistical Analysis Plan for PDC-1421 "Final"  Protocol Version: 2.3 SAP Version: 20180626 01

### 8. DATA HANDLING PROCEDURE

# 8.1 Coding System

The MedDRA system (version 20.0) is used to code adverse events.

Concomitant medication will be coded via WHODRUG.

General medical history term will be coded via ICD-10 coding system

# 8.2 Data Storage and Analysis

All data are stored in the VCROCTIS system.

Statistical evaluation will be performed using SAS 9.4 (SAS-Institute Inc., Cary, NC).

Project No. BLI-1005-002 Statistical Analysis Plan for PDC-1421

### **"Final"**  Protocol Version: 2.3 SAP Version: 20180626 01

## 9. STUDY SUBJECTS

# 9.1 Disposition of Subjects

The number and percentage of randomized subject no. and analysis population will be tabulated by center and treatment.

## 9.2 Withdrawal of Subjects

Frequency table of the reasons for subject withdraw from study will be presented by center and treatment.

### 9.3 Protocol Deviations

Protocol deviations will be listed and will be tabulated by center and treatment.

Project No. BLI-1005-002 Statistical Analysis Plan for PDC-1421 **"Final"**  Protocol Version: 2.3 SAP Version: 20180626 01

## 10. REFERENCE LIST

Clenn A. Walker, Common Statistical Methods for Clinical Research with SAS® Examples, 2nd edition, Cary, NC, SAS Institute Inc., 2002

Shein-Chung Chow, Jen-pei Liu, Design and Analysis of Clinical Trials, John Wiley & Sons, Inc., 1998

Project No. BLI-1005-002 Statistical Analysis Plan for PDC-1421 **"Final"**  Protocol Version: 2.3 SAP Version: 20180626 01

## 11. APPENDICES

## 11.1 Normal Ranges For Laboratory Variables

Will be listed in data listings

# 11.2 Table of Contents (TOC) for Tables, Figures and Listing

Refer to section 14 and 16.2 in clinical study report

No further SAP amendment will be required for the deviation of TOC when the changes are still complied with the main text SAP.

### 11.3 Mock-up tables

Refer to attachment "MUT\_BOLPDCA20141117\_20180626\_01\_final\_20190611.pdf"

### 11.4 Version Control Information of SAP

| Document | Version | Approved date |
|----------|-------------|---------------|
| Final | 20180626_00 | Apr-19-2019 |
| Final | 20180626_01 | June-14-2019 |

Project No. BLI-1005-002 Statistical Analysis Plan for PDC-1421 "Final"  Protocol Version: 2.3 SAP Version: 20180626\_01

## 11.5 Contents of Amendment of SAP

| Page | Before | Page | Content after modification |
|---|---|---|---|
| | version: 00 | | Version: 01 |
| 20~ 21 | 6.4 Analysis of Efficacy Results of efficacy will be presented with descriptive statistics (i.e. sample size, number of missing data, mean, 95% confidence interval of mean, median, standard deviation, interquartile range, maximum and minimum) for continuous parameters by part, visit, and treatment. | 20~<br>21 | 6.4 Analysis of Efficacy Results of efficacy will be presented with descriptive statistics (i.e. sample size, number of missing data, mean, 95% confidence interval of mean, median, standard deviation, inter- quartile range, maximum and minimum) for continuous parameters by part, visit, and treatment. Line charts of all efficacy outcomes will be generated and presented as mean and standard deviation. |
| 22 | Definition of partial responderpartial responder are defined as participants with at least 25% and no more than 50% decrease in total score from baseline) and the 95% confidence interval (CI) will be computed. | 22 | Definition of partial responderpartial responders are defined as participants with at least 25% and no more than 50% decrease in total score from baseline). |
| 22 | 6.5.1 Adverse events (AEs) For TEAE, incidence tables of severity, action taken, relationship to study drug, outcome and serious AE or not will be presented by part, center, and treatment. | 22 | 6.5.1 Adverse events (AEs) For TEAE, incidence tables of severity, action taken, relationship to study drug, outcome and serious AE or not will be presented by part, center, preferred term and treatment. The frequency distribution of severity, action taken, relationship to study drug, and outcome of all AE events will be presented by part, center, and treatment. |
| 23 | 6.5.4 Physical Examination (PE) Only when abnormality is recorded, the corresponding body system will be analyzed and reported using a transition table. The type of transition includes normal -> normal, normal -> abnormal, abnormal -> abnormal, and abnormal-> normal for each body system from baseline (Visit 2). | 23 | 6.5.4 Physical Examination (PE) The corresponding body system will be analyzed and reported using a transition table. The type of transition includes no change, change to normal, change to non-clinical significance, (NCS), change to clinical significance (CS) for each body system from baseline (Visit 2). |
| 23 | 6.5.5 Vital Signs Descriptive statistics of net changes in vital signs including systolic and diastolic blood pressure, heart rate and | 23 | 6.5.5 Vital Signs Descriptive statistics of net changes in vital signs including systolic and diastolic blood pressure, heart rate and |

Sponsor: BioLite, Inc.

Project No. BLI-1005-002 Statistical Analysis Plan for PDC-1421

"Final"  Protocol Version: 2.3 SAP Version: 20180626\_01

| | body temperature will be presented by part, center, visit, and treatment. | | body temperature will be presented by part, center, visit, and treatment. Results of clinical significance with regard to vital sign will be summarized with frequency and percentage. |
|---|---|---|---|
| 23 | 6.5.6 ECG Frequency table and change in ECG result will be summarized by part, center, visit and treatment. The transition of ECG is define as following 4 groups: normal -> normal, normal -> abnormal, abnormal -> abnormal, and abnormal-> normal. | 23 | 6.5.6 ECG Frequency table and change in ECG result will be summarized by part, center, visit and treatment. The transition of ECG is define as following 4 groups: no change, change to normal, change to non-clinical significance, (NCS), change to clinical significance (CS). |
| 30 | 11.3 Mock-up tables Refer to attachment "MUT_BOLPDCA20141117_20180626_ 00_final20190411.pdf" | 30 | 11.3 Mock-up tables Refer to attachment "MUT_BOLPDCA20141117_20180626 _01_final_20190611.pdf" |